CLINICAL TRIAL: NCT00779142
Title: Evaluation of the Utility of Intravitreal Methotrexate in Patients With Recalcitrant Diabetic Macular Edema in an Open Label, Nonrandomized, Uncontrolled, Interventional Pilot Trial
Brief Title: Utility of Intravitreal Methotrexate in Diabetic Macular Edema Resistant to Conventional Therapies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recent research indicates Lucentis to be an effictive treatment
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5865 Methotrexate
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-11

CONDITIONS: Diabetic Macular Edema
Keywords: resistant diabetic macular edema
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate 25mg/ml (Other): Methotrexate intravenous 25mg/ml: Methotrexate intravenous 25mg/ml delivered once or twice (based on the therapeutic response) over a period of 2 months maximum. Total dosage 400ug in each dose to subjects with diabetic macular edema resistant to conventional therapies.
  Interventions: Drug: Methotrexate intravenous 25mg/ml

INTERVENTIONS:
Drug: Methotrexate intravenous 25mg/ml — Methotrexate intravenous 25mg/ml delivered once or twice (based on the therapeutic response) over a period of 2 months maximum. Total dosage 400ug in each dose. Statistical analysis would not be applicable in this small sample.
  Other Names: Methotrexate

SUMMARY:
It is well known that blindness is one of the most feared disabilities expressed by patients in the United States. Estimates of the economic impact of visual disability in the current population exceed 30 million US dollars in this country alone. The reasons for this figure are many; however age related macular degeneration (ARMD), diabetic retinopathy, glaucoma and uveitis are responsible for the majority of permanent visual disability and hence the costs in both quality of life and placing an economic burden on society. Research that may help reverse various abnormal biological responses that lead to or worsen clinical manifestations of diabetic retinopathy would be valuable.

DETAILED DESCRIPTION:
The most common reason for decreased vision in diabetic retinopathy is macular edema. Current approaches to macular edema include FDA approved interventions such as laser and better underlying control of the disease and co morbid conditions. 'Off label' interventions include intravitreal triamcinolone and bevacizumab, both of which have been demonstrated to be efficacious; at least in the short term (weeks) but carry significant risks. Surgical approaches are still controversial and have not shown long term benefits. Unfortunately, there are subsets of patients resistant to any of the above therapies. Intravitreal therapies utilizing methotrexate 400 ug (MTX) have been used for other ophthalmologic conditions associated with inflammation driven macular edema. bevacizumab an anti VEGF agent has been utilized in diseases other than macular degeneration with a favorable effect. It is known that certain similar inflammatory mediators play a role in diabetic macular edema. It would be logical to evaluate the efficacy of MTX an anti inflammatory anti metabolite at low concentrations in diabetic patients with macular edema who have failed conventional FDA approved and well studied off label therapies that involve laser and/or intravitreal drugs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) with clinically significant macular edema (CSME) with visual acuity less than 20/60 to Hand motion in the study eye.
* Patients should have persistent CSME three months after laser therapy or three months after intraocular injection of Avastin or triamcinolone. These interventions could be multiple or combined.
* Optical coherence tomography (OCT) scan demonstrating more than 275 microns retinal thickness in central subfield of study eye.
* Ability to understand study instructions, interventions and potential complications.
* History of reasonably controlled Diabetes mellitus (DM), ≤ 8.5HbA1c that has been evaluated in the last 3 months.
* Ability to undergo contraceptive protection during and 3 months after intraocular injections.
* Clear demonstration (in female patients) of commitment to avoid pregnancy and a negative urine pregnancy test at baseline for women of childbearing potential.
* Clear understanding of teratogenic potential of MTX.

Exclusion Criteria:

* History of allergy to MTX.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition.
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, epiretinal membrane, etc.).
* An eye treated for Glaucoma
* Eyes that underwent vitrectomy
* History of intraocular malignancies.
* Intraocular surgery with the prior 3 months.
* Recent significant change in diabetic medications.
* Insulin usage less than a year.
* Life threatening co morbidities such as cancer under therapy.
* Use of oral, intravenous, periocular or intraocular corticosteroids (steroids) in prior 3 months.
* Liver function that exceeds three times the upper limit of normal at baseline, or within 6 weeks of that appointment.
* Pregnant females.
* Vitreous hemorrhage (active) in study eye
* Anticipation of the need for laser pan retinal photocoagulation in the next 6 months.
* Media opacities
* Herpetic disease of cornea
* Corneal dystrophy with significant corneal edema.
* Any major surgery within the last 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shree K Kurup, MD, Principal Investigator — Wake Forest Baptist Health Eye Center
Locations (1):
- Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rein DB, Zhang P, Wirth KE, Lee PP, Hoerger TJ, McCall N, Klein R, Tielsch JM, Vijan S, Saaddine J. The economic burden of major adult visual disorders in the United States. Arch Ophthalmol. 2006 Dec;124(12):1754-60. doi: 10.1001/archopht.124.12.1754. PMID 17159036
- [Background] Shimura M, Nakazawa T, Yasuda K, Shiono T, Iida T, Sakamoto T, Nishida K. Comparative therapy evaluation of intravitreal bevacizumab and triamcinolone acetonide on persistent diffuse diabetic macular edema. Am J Ophthalmol. 2008 May;145(5):854-61. doi: 10.1016/j.ajo.2007.12.031. Epub 2008 Mar 6. PMID 18328456
- [Background] Vasconcelos-Santos DV, Nehemy PG, Schachat AP, Nehemy MB. Secondary ocular hypertension after intravitreal injection of 4 mg of triamcinolone acetonide: incidence and risk factors. Retina. 2008 Apr;28(4):573-80. doi: 10.1097/IAE.0b013e31816079e8. PMID 18398360
- [Background] Hartley KL, Smiddy WE, Flynn HW Jr, Murray TG. Pars plana vitrectomy with internal limiting membrane peeling for diabetic macular edema. Retina. 2008 Mar;28(3):410-9. doi: 10.1097/IAE.0b013e31816102f2. PMID 18327132
- [Background] Hardwig PW, Pulido JS, Erie JC, Baratz KH, Buettner H. Intraocular methotrexate in ocular diseases other than primary central nervous system lymphoma. Am J Ophthalmol. 2006 Nov;142(5):883-5. doi: 10.1016/j.ajo.2006.06.002. PMID 17056381
- [Background] Ghajarnia M, Kurup S, Eller A. The therapeutic effects of intravitreal bevacizumab in a patient with recalcitrant idiopathic polypoidal choroidal vasculopathy. Semin Ophthalmol. 2007 Apr-Jun;22(2):127-31. doi: 10.1080/08820530701421635. PMID 17564935

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate 25mg/ml: Methotrexate intravenous 25mg/ml delivered once or twice (based on the therapeutic response) over a period of 2 months maximum. Total dosage 400ug in each dose. Statistical analysis would not be applicable in this small sample.
  Methotrexate intravenous 25mg/ml: Methotrexate intravenous 25mg/ml delivered once or twice (based on the therapeutic response) over a period of 2 months maximum. Total dosage 400ug in each dose. Statistical analysis would not be applicable in this small sample.
Period: Overall Study
Arm/Group | Methotrexate 25mg/ml
Started | 5 (5 patients signed consent and were screened.)
Completed | 2 (Only 2 patients were actually enrolled.)
Not Completed | 3
Not completed — Screen Failures | 3

BASELINE CHARACTERISTICS:
Population: Patients with Recalcitrant Diabetic Macular Edema
Groups:
- Methotrexate 25mg/ml: Methotrexate intravenous 25mg/ml delivered once or twice (based on the therapeutic response) over a period of 2 months maximum. Total dosage 400ug in each dose. Statistical analysis would not be applicable in this small sample.
Arm/Group | Methotrexate 25mg/ml
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (19.05781)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: 30% Decrease in One Subfield Thickness on Optical Coherence Tomography (OCT) 4 Weeks After the Last Intraocular Injection
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Methotrexate 25mg/ml
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Number of Participants With Increase in Visual Acuity (VA) Two Lines or More at the End of One Month After the Last Intraocular Injection
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate 25mg/ml
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Secondary Would be Significant Clinical Improvement (Judged at the Slit Lamp Exam Using a 90D Lens) in Macular Edema at the End of One Month After the Last Intraocular Injection.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate 25mg/ml
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Arm/Group | Methotrexate 25mg/ml
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes